CLINICAL TRIAL: NCT02168660
Title: Normalization of Vitamin D Levels and Its Effect on Glucose Homeostasis in Obese Youth
Brief Title: Correction of Vitamin D Levels and Its Effect on Insulin Resistance and Weight Gain in Obese Youth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Perrin C White, MD (Other)
Responsible Party: Sponsor-Investigator, Perrin C White, MD, Professor of Pediatrics, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UT092010-217
Record Dates: First submitted 2014-06-17; First posted 2014-06-20 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Obesity; Insulin Resistance; Vitamin D Deficiency
Keywords: Obesity; Insulin Resistance; Vitamin D Deficiency; Children; Adolescents
MeSH Terms: conditions — Obesity; Insulin Resistance; Vitamin D Deficiency | interventions — Cholecalciferol; Calcifediol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Group (Active Comparator): Standard vitamin D3 dose as per IOM (Institute of Medicine) recommendations; actual dose will be 5000 IU per week, which is just slightly higher than the IOM recommendation of 600 IU per day. Length of time proposed to be 4 months at 5000 IU D3 per week. End of study measures at 4 months to be HOMA-IR, BMI Z score, 25-OHD level.
  Interventions: Drug: Vitamin D3
- Low-Normal Group (Experimental): Initial D3 dose will be 30,000 IU per week; at 6 week intervals serum D3 levels will be checked, and dose adjustments made to reach target 25-OHD level of between 30-50 ng/mL (inclusive). Once within target, D3 dose will be continued for 4 months, and end of study measurements done (HOMA-IR, BMI Z score, 25-OHD level).
  Interventions: Drug: Vitamin D3
- High-Normal Group (Experimental): Initial D3 dose will be 60,000 IU/week; at 6 week intervals 25-OHD levels will be done, and dose adjustments made to achieve target level of 40-60 ng/mL (inclusive). Once within target range, D3 dose will be continued for 4 months, and end of study measures obtained (HOMA-IR, BMI Z score, 25-OHD level).
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3, liquid formulation, 5000 IU/mL.
  Other Names: calcidiol

SUMMARY:
Vitamin D deficiency is extremely common in obese youth. In our obese population followed in the Endocrinology clinic at Children's Medical Center Dallas, vitamin D levels were inversely correlated with a measure of insulin resistance. We propose to show that correction of vitamin D levels in obese children and adolescents improves their insulin sensitivity. Obese youth presenting to the Center for Obesity and its Consequences on Health (COACH) clinic will be randomized to receive either the most recent Institute of Medicine (IOM) recommendations of minimum D3 dose of 600 IU/day (1), or receive higher doses of D3 such that the blood levels of vitamin D will be brought to a target level in either the low part or high part of the normal range. The goal is to determine if correction of vitamin D deficiency will improve insulin sensitivity in this group. Secondary goals include determining whether correction of vitamin D deficiency in obese adolescents and children results in less weight gain, and determining the amount of D3 required to correct vitamin D levels in this population.

Our specific hypotheses are as follows:

Hypothesis #1 Obese youth treated with Vitamin D3 who achieve low-normal 25-hydroxyvitamin D3 (OHD) levels (30-50 ng/mL) or high-normal 25-OHD levels (60-80 ng/mL) will have improved insulin resistance, as measured by Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), compared to those individuals with deficient 25-OHD levels (< 30 ng/mL).

Hypothesis #2 Subjects with a higher BMI will have higher Vitamin D dose requirements than current IOM recommendations of 600 IU/day and will take a longer period of time to reach target 25-OHD levels.

Hypothesis #3 Subjects with normal 25-OHD levels will demonstrate less weight gain compared to subjects on the control arm.

DETAILED DESCRIPTION:
Concise Summary of Project: The proposed study is a prospective, unblinded dose-ranging trial to examine in obese youth 1) the effect of correcting Vitamin D (Vit D) deficiency on insulin resistance, 2) the effect of correcting Vit D deficiency on weight gain, and 3) the amount of Vit D3 required to achieve Vit D sufficiency in obese adolescents. Subjects will be recruited from obese children and adolescents aged 6 to 17 years presenting to the COACH clinic, a referral clinic for obese children at Children's Medical Center of Dallas. Approximately 1300 new patients are seen in the COACH clinic each year. Ethnicity will be self-assigned as African-American, Caucasian, Hispanic, or Other. The ethnic makeup of the COACH clinic over the last 20 months was as follows: African-American 25%, Caucasian 19.5%, Hispanic 52%, and Other 3.5%.

As per standard practice in the COACH clinic, a height (cm), weight (kg), and blood pressure will be obtained, and body mass index (kg/m2) calculated for each patient. Fasting total cholesterol, LDL, HDL, triglyceride, 25-OHD, Hemoglobin A1c (A1c), and fasting insulin will be obtained, and an Oral Glucose Tolerance Test (OGTT) performed. The baseline estimate of insulin sensitivity is calculated from the fasting insulin and glucose values, and reported as the HOMA-IR. After Informed Consent has been obtained, participants will be randomized to either the Control group (5000 IU/wk), the Low-normal 25-OHD group (target 25-OHD 30-50 ng/mL), or the High-normal 25-OHD group (target 25-OHD 60-80 ng/mL). A 25-OHD < 25 ng/mL will be confirmed. These groups will be matched for age (6-12 years versus 13-17 years) and ethnicity (Caucasian versus African-American verus Hispanic). Approximately 60 patients will be recruited for each group. Subject participation will continue until Vit D sufficiency has been documented for 4 consecutive months, at which point the fasting insulin and glucose values will be repeated for calculation of HOMA-IR and assessment of insulin sensitivity, and amount of weight gain will be measured.

ELIGIBILITY:
Inclusion Criteria:

* age 6-17 years
* BMI > 95% for age
* serum 25-OH D level < or + to 25 ng/mL

Exclusion Criteria:

* BMI < 95% for age
* serum 25-OH D level > 25 ng/mL
* current Vitamin D supplementation > 400 IU/day
* anti-convulsant therapy, anti-hypertensive therapy, lipid lowering medication
* any medications that affect glucose metabolism (e.g., metformin, insulin)
* daily glucocorticoid therapy
* diabetes
* any disorders of bone or calcium metabolism
* hepatic or renal disease
* any malabsorptive disorder
* baseline serum Calcium > 11 ng/dL (> 2 SD above the mean)
* any genetic disorder that predisposes to obesity (e.g., Prader Willi
* hypothalamic obesity

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 109 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2015-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele R Hutchison, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Olson ML, Maalouf NM, Oden JD, White PC, Hutchison MR. Vitamin D deficiency in obese children and its relationship to glucose homeostasis. J Clin Endocrinol Metab. 2012 Jan;97(1):279-85. doi: 10.1210/jc.2011-1507. Epub 2011 Nov 9. PMID 22072738
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827
- [Background] Mansbach JM, Ginde AA, Camargo CA Jr. Serum 25-hydroxyvitamin D levels among US children aged 1 to 11 years: do children need more vitamin D? Pediatrics. 2009 Nov;124(5):1404-10. doi: 10.1542/peds.2008-2041. PMID 19951983
- [Background] Rajakumar K, Fernstrom JD, Holick MF, Janosky JE, Greenspan SL. Vitamin D status and response to Vitamin D(3) in obese vs. non-obese African American children. Obesity (Silver Spring). 2008 Jan;16(1):90-5. doi: 10.1038/oby.2007.23. PMID 18223618
- [Background] Bischoff-Ferrari HA, Giovannucci E, Willett WC, Dietrich T, Dawson-Hughes B. Estimation of optimal serum concentrations of 25-hydroxyvitamin D for multiple health outcomes. Am J Clin Nutr. 2006 Jul;84(1):18-28. doi: 10.1093/ajcn/84.1.18. PMID 16825677
- [Background] Nagpal J, Pande JN, Bhartia A. A double-blind, randomized, placebo-controlled trial of the short-term effect of vitamin D3 supplementation on insulin sensitivity in apparently healthy, middle-aged, centrally obese men. Diabet Med. 2009 Jan;26(1):19-27. doi: 10.1111/j.1464-5491.2008.02636.x. PMID 19125756
- [Background] von Hurst PR, Stonehouse W, Coad J. Vitamin D supplementation reduces insulin resistance in South Asian women living in New Zealand who are insulin resistant and vitamin D deficient - a randomised, placebo-controlled trial. Br J Nutr. 2010 Feb;103(4):549-55. doi: 10.1017/S0007114509992017. Epub 2009 Sep 28. PMID 19781131
- [Background] Alemzadeh R, Kichler J, Babar G, Calhoun M. Hypovitaminosis D in obese children and adolescents: relationship with adiposity, insulin sensitivity, ethnicity, and season. Metabolism. 2008 Feb;57(2):183-91. doi: 10.1016/j.metabol.2007.08.023. PMID 18191047
- [Background] Maalouf J, Nabulsi M, Vieth R, Kimball S, El-Rassi R, Mahfoud Z, El-Hajj Fuleihan G. Short- and long-term safety of weekly high-dose vitamin D3 supplementation in school children. J Clin Endocrinol Metab. 2008 Jul;93(7):2693-701. doi: 10.1210/jc.2007-2530. Epub 2008 Apr 29. PMID 18445674

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Standard vitamin D3 dose as per IOM (Institute of Medicine) recommendations; actual dose will be 5000 IU per week, which is just slightly higher than the IOM recommendation of 600 IU per day. Length of time proposed to be 4 months at 5000 IU D3 per week. End of study measures at 4 months to be HOMA-IR, BMI Z score, 25-OH D level.
  Vitamin D3: Vitamin D3, liquid formulation, 5000 IU/mL.
- High-Normal Group: Initial D3 dose will be 60,000 IU/week; at 6 week intervals 25-OHD levels will be done, and dose adjustments made to achieve target level of 40-60 ng/mL (inclusive). Once within target range, De3 dose will be continued for 4 months, and end of study measures obtained (HOMA-IR, BMI Z score, 25-OHD level).
  Vitamin D3: Vitamin D3, liquid formulation, 5000 IU/mL.
Period: Overall Study
Arm/Group | Control Group | Low-Normal Group | High-Normal Group
Started | 38 | 35 | 36
Completed | 22 | 18 | 21
Not Completed | 16 | 17 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Low-Normal Group | High-Normal Group | Total
Number analyzed (Participants) | 22 | 18 | 21 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 18 | 21 | 61
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 12 [10 to 14] | 12 [11 to 13] | 13 [11 to 14] | 12 [11 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 10 | 29
  Male | 13 | 8 | 11 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 16 | 15 | 48
  Not Hispanic or Latino | 5 | 2 | 6 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 5 | 8
  White | 19 | 16 | 16 | 51
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 22 | 18 | 21 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in HOMA-IR
Description: Change in HOMA-IR from initial visit to end-of-study visit; i.e., the value at the later time point minus the value at the earlier time point. HOMA-IR= Fasting insulin (mIU/ml) x Fasting glucose (mg/dl) / 405.
Time Frame: 4-12 mo after randomization (4 months after target 25-hydroxyvitamin D level is reached).
Population: Beginning and ending anthropometric data were available within the specified time limits on 61 subjects and 25-hydroxyvitamin D3 (25-OHD) levels on 45. Corresponding insulin and glucose data (allowing calculation of HOMA-IR) were available on only 26 subjects, mainly because many 25-OHD levels were obtained when subjects were not fasting.
Measure: Median (Inter-Quartile Range); unit: HOMA-IR score
Arm/Group | Control Group | Low-Normal Group | High-Normal Group
Number analyzed (Participants) | 7 | 11 | 8
HOMA-IR score | 0 [-1.8 to 1.4] | -1.5 [-3.9 to 0.9] | -1.7 [-4.3 to -0.3]

2. Secondary Outcome: Time to Normalization of Vit D Level Versus BMI Z Score
Description: The time required to reach a normal Vitamin D level (> 30) versus BMI Z score at each vitamin D3 dose; OR vitamin D level at 6 weeks versus BMI Z score at each starting vitamin D3 dose.
Time Frame: 1 to 12 months
Population: Timing of sample collections was too irregular to permit analysis.
Arm/Group | Control Group | Low-Normal Group | High-Normal Group
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change in BMI Z-score
Description: The change in BMI z-score from baseline to end-of-study visit; i.e., the value at the later time point minus the value at the earlier time point.
  The BMI Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched children). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population.
Time Frame: 4-12 mo after randomization (4 months after target 25-hydroxyvitamin D level is reached).
Measure: Median (Inter-Quartile Range); unit: z-score
Groups:
- Control Group: Standard vitamin D3 dose as per IOM (Institute of Medicine) recommendations; actual dose will be 5000 IU per week, which is just slightly higher than the IOM recommendation of 600 IU per day. Length of time proposed to be 4 months at 5000 IU D3 per week. End of study measures at 4 months to be HOMA-IR, BMI z-score, 25-OH D level.
  Vitamin D3: Vitamin D3, liquid formulation, 5000 IU/mL.
- Low-Normal Group: Initial D3 dose will be 30,000 IU per week; at 6 week intervals serum D3 levels will be checked, and dose adjustments made to reach target 25-OHD level of between 30-50 ng/mL (inclusive). Once within target, D3 dose will be continued for 4 months, and end of study measurements done (HOMA-IR, BMI z-score, 25-OHD level).
  Vitamin D3: Vitamin D3, liquid formulation, 5000 IU/mL.
- High-Normal Group: Initial D3 dose will be 60,000 IU/week; at 6 week intervals 25-OHD levels will be done, and dose adjustments made to achieve target level of 40-60 ng/mL (inclusive). Once within target range, De3 dose will be continued for 4 months, and end of study measures obtained (HOMA-IR, BMI z-score, 25-OHD level).
  Vitamin D3: Vitamin D3, liquid formulation, 5000 IU/mL.
Arm/Group | Control Group | Low-Normal Group | High-Normal Group
Number analyzed (Participants) | 22 | 18 | 21
z-score | 0.03 [-0.04 to 0.07] | -0.07 [-0.11 to -0.03] | -0.03 [-0.12 to 0.0]

ADVERSE EVENTS:
Arm/Group | Control Group | Low-Normal Group | High-Normal Group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18 | 0/21
Other Adverse Events (participants affected / at risk) | 0/22 | 1/18 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=22) | Low-Normal Group (N=18) | High-Normal Group (N=21)
abdominal pain (Gastrointestinal disorders) | 0 | 1 (1) | 0

LIMITATIONS AND CAVEATS:
Because of poor subject retention, there were insufficient outcome data to allow hypothesis testing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes